CLINICAL TRIAL: NCT03935243
Title: Efficacy of Equine Assisted Therapy on Psychosocial Functioning, Negative Symptoms and Quality of Life in Patients With Schizophrenia: a Prospective, Randomised and Controlled Study
Brief Title: Efficacy of Equine Assisted Therapy on Negative Symptoms in Patients With Schizophrenia
Acronym: STABLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-STABLE
Record Dates: First submitted 2019-04-11; First posted 2019-05-02 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Animal Assisted Therapy
MeSH Terms: interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- equine assisted therapy (Experimental): In the active intervention phase, patients participate twice a week in a equine assisted group therapy, while during the control phase they participate twice a week in a group that includes a non-specific and general activity program. After 15 therapy units in a study phase, the subjects will complete the 15 units of the other study phase (within-subject-design). All participants complete both study phases, with the order being randomized.
  Interventions: Behavioral: equine assisted therapy
- activating control phase (Active Comparator): In the present study, the interventions in the control phase are based on the sub-program "Social Skills" of the Integrated Psychological Treatment Program (IPT) for schizophrenic patients (Brenner et al., 1994, Roder et al., 1988, 2002).
  Interventions: Behavioral: activating control phase

INTERVENTIONS:
Behavioral: equine assisted therapy — The equine assisted group therapy is carried out by a riding therapist (nurse psychiatry HF, certified riding therapist SG-TR). There is a detailed plan for the PT.
  Arms: equine assisted therapy
Behavioral: activating control phase — The control phase includes a generally activating employment offer, such as board games, light physical activations, roundtables and artistic design.
  Arms: activating control phase

SUMMARY:
The main object of this study is to evaluate the efficacy of equine assisted therapy on substantial and so far unsatisfactorily treatable symptom complexes in patients with schizophrenia.

DETAILED DESCRIPTION:
The clinical picture in schizophrenia involves changes in perception, cognition, and affect such as delusions, hallucinations, and disorganized thinking and disorders of attention, memory, and executive thinking. A clinical differentiation, which is widespread in practice, divides the psychopathological disorders of schizophrenic patients in the clinical core areas into positive and negative symptoms.

The term negative symptoms was introduced by Hughlings-Jackson, who made the distinction between florid-psychotic or positive symptoms and "defect" or negative symptoms. The term "positive symptoms" usually includes delusions, hallucinations and formal thinking disorders. The latter are often explained in recent research tradition as a separate "disorganization syndrome". Negative symptoms also appear in the context of other psychiatric and neurological disorders, for example in patients with depression, Parkinson's and craniocerebral traumas.

Negative symptoms, according to Frith and Done, essentially signify a "deficit of willed action" or, more generally, a pathological deficit of activity and reactivity. To establish a border between idiopathic, i.e. primarily due to schizophrenia, outlasting ("trait") negative symptoms and secondary, temporary ("state") negative symptoms Carpenter and colleagues introduced the concept of the deficit vs. non-deficit form of schizophrenia. Negative symptoms constituting the deficit syndrome include affective flattening, limited emotional range, loss of interest, speech depletion, diminished purposefulness, and social listlessness. These symptoms are considered to be primary negative symptoms if they persist beyond the onset of an acute psychotic episode and have been established by differential diagnosis that they are not or at least not entirely secondary to the presence of depression, the side effects of antipsychotic treatment or other circumstances. While primary negative symptoms are currently largely immune to any type of treatment, secondary negative symptoms may remit spontaneously or after appropriate treatment.

Men are more frequently and stronger affected by negative symptoms than women. Also, the negative symptoms manifest themselves earlier in the course of the disease and are associated with stronger cognitive impairments than in women. However, the extent of men's deficits varies little during further psychotic episodes, while women tend to have a progressive profile. Recruitment for the current study will take into account the prevalence.

The positive symptoms can be treated very effectively with medication and stabilization can usually be achieved within a few weeks. On the other hand, the negative symptoms are very difficult to influence with medication. Ideally, modern integrative psychiatric treatment concepts therefore incorporate a combination of pharmacological, psychotherapeutic and psychosocial treatment strategies adapted to the specific symptom constellation and the particular needs and deficiencies of the individual patient.

In recent years, a wide variety of treatments (e.g. transcranial magnetic stimulation or psychosocial treatment options) have been used to improve the negative symptoms in schizophrenic patients, but treatment success has remained low. Thus, the results of existing studies on TMS and rTMS are also controversial. There are some studies in which positive effects were found on the psychpathology for example, whereas other studies could not find any significant positive effects of rTMS in schizophrenia patients.

Another applied intervention that has been established for many years in a wide variety of mental illnesses is animal assisted therapy. This is used for example in children with autism, patients with anxiety disorders or depression, but also in schizophrenic patients. The effects of animal assisted therapy are versatile. For example, improvements in autistic symptoms, emotional well-being, self-esteem, self-determination, depressive symptoms, positive and negative symptoms in schizophrenics or improvement in quality of life were found.

In studies that explicitly examined the effects of animal assisted therapy on schizophrenic patients, several positive outcomes have been reported. Maujean and colleagues found in their meta-analysis positive effects of animal assisted therapy on social contact, positive and negative symptoms, and the quality of life in terms of interpersonal relationships. Barak and colleagues investigated in their study how animal assisted therapy affects older schizophrenic patients and found a significant improvement on the Social Adaptive Functioning (SAFE) scale with a focus on the social function subscale. Furthermore, positive effects on the activities of everyday life and general well-being were found. There were several studies which assessed the PANSS (Positive and Negative Syndrome Scale) and found a significant improvement in the negative symptoms due to animal assisted therapy. In addition, a reduction of the cortisol level was noted and the adherence in the therapy group compared to the control group was significantly higher. Furthermore, a constant remission of the disease as well as a lower hospitalization of the patients were reported. One study, in addition to the PANSS, the Living Skills Profile (LSP) and the World Health Organization Quality of Life Assessment (WHOQOL-BREF) letter were included and a significant effects on both scales was found as well. In another meta-analysis conducted by Jormfeldt and Carlsson in 2018, six months after the last intervention, positive effects continued to be found at follow-up. Participants in animal assisted therapy reported benefits at the psychosocial level, such as increased self-efficacy and self-esteem, social stimulation, and new skills that could be transferred to other areas of life. In summary, there is already evidence for the efficacy of animal assisted therapy on the negative symptoms, psychosocial functioning and quality of life of schizophrenic patients, which should be further supported in the controlled setting as part of the planned study.

Appropriate conceptualization is essential for the development of suitable treatment methods for the negative symptoms of schizophrenic patients. However, the concept of negative symptoms has changed significantly since the development of the standard instruments SANS and PANSS, and for a long time there was no clear consensus on the construct of negative symptoms.

In their 2014 review, Marder & Kirkpatrick juxtaposed the standard instruments SANS and PANSS with newer gauges designed to assess negative symptoms. As one of the first scales designed exclusively for the detection of negative symptoms in schizophrenic patients, the SANS has played a key role in the holistic study of schizophrenia. However, Marder & Kirkpatrick argue that the SANS contains items that are unlikely to be part of the negative symptoms (inappropriate affect & impaired attention). These items have also often been omitted by researchers in recent years when using the SANS. Furthermore, more recent studies suggest that it would be useful to distinguish between the anticipatory and the consumptive aspect of anhedonia, as the patients do have some limitations in the first, but this does not seem to be the case with the latter. At a National Consensus Meeting held by the NIMH (National Institut for Mental Health), negative symptom domains were identified that are inconsistent with the five subscales of the SANS or the five factors of the PANSS. The fixed domains are dulled affect, alogy, asociality, anhedonia, and avolition. A scale used to record the negative symptoms should accordingly only contain items that belong to the above-mentioned areas. Another issue is that the meter should be able to detect changes in the symptoms. In addition, it should be short and internationally applicable (easy to translate and transferable to different cultures). Finally, a measurement tool should have psychometric properties such as inter-rater reliability, internal consistency, test-retest reliability, and content, convergence, and discriminant validity.

Under these conditions, the BNSS emerged. This short scale for detecting negative symptoms in schizophrenic patients consists of 13 items and can be collected within 15 minutes. It was important to the authors of the scale to distinguish between the anticipatory and consumptive aspects of anhedonia, as well as between experience and behavior. The BNSS showed excellent inter-rater and test-retest reliability, as well as good vailidity in comparison with other scales, as shown in psychometric studies. Furthermore, it could be shown that the scale has an inverse correlation with a measure of the functional level and the MATRICS Consensus Battery. An additional important point is that the BNSS correlates only marginally with masses of positive symptoms, anxiety, and depression. For these reasons, the BNSS should also be used in the planned study. In addition, the further development of objective measuring instruments for the collection of negative symptoms in the study by examining the application of acoustic analysis and the concept of the voice should explain changes in schizophrenia as a correlate of negative symptoms.

Other target variables of the study will be the PSP scale (Personal and Social Performance Scale) and the S-QoL (Quality of Life Questionnaire in Schizophrenia). The PSP was designed out of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) with the goal to develop a scale that can quickly and validly capture the personal and psychosocial functioning of patients. Among the advantages of the PSP over other scales such as the SOFAS or the GAF (Global Assessment of Functioning), is the fact that the professional, social and personal functioning are operationalized in more detail, since there is no mixing of psychopathological symptoms and psychosocial aspects. Furthermore, the four subscales of the PSP, which are initially collected in order to then form a total score, give a higher information value than is the case with the SOFAS or the GAF . In addition, initial studies on the PSP have shown that the scale has high validity and reliability values. The PSP is a third-party assessment and, as already mentioned, contains four subscales whose items are queried on a 6 point scale. From the assessments of the four subscales, an overall score is then formed, ranging from 0-100 and subdivided into 10 intervals. To simplify the survey, Schaub and Juckel have developed an interview guide for the German version of the PSP.

As mentioned above, the recovery and improvement of psychosocial functioning have become increasingly the focus of treatment efforts in recent years. In this context, the quality of life of patients was often examined. As a secondary target variable, therefore, an instrument for assessing the subjective quality of life should also be used in the planned study. Despite the large number of life-quality assessment tools validated or specifically developed for schizophrenic patients in recent years, there is no clear consensus on which survey instrument to use. The selection should therefore focus on the concrete conceptualization of the instrument, the question and the applicability of the population to be examined in the existing setting. In the present study, the Quality of Life Questionnaire is to be applied in schizophrenia (S-QoL). It uses 41 items to record 8 subscales of the quality of life such as well-being, self-esteem, resilience and autonomy. The S-QoL is a self-assessment tool and its application takes 15 minutes.

The present study STABLE is planned with inpatients at the Psychiatric University Clinic, Department of Forensic Psychiatry, Center for Inpatient Forensic Therapy Rheinau. In the active control phase, a WHO-recommended psychosocial intervention for the treatment of schizophrenia, the training of everyday activities and self-employment (board games, everyday skills, etc.) is used. In terms of content, the training of everyday activities is based on the sub-program "Social Skills" of the IPT (Integrated Psychological Therapy Program).

The study complies with the European Mental Health Action Plan 2013-2020.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (ICD-10: F20.0-20.3, F20.5)
* men or female patients (older than 18 years of age)
* written informed consent

Exclusion Criteria:

* acute risk of harming oneself or others
* severe manifest allergies
* medically uncontrolled epilepsy
* Significant side effects of medication (blood pressure fluctuations with dizziness, movement-limiting Parkinson's disease, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changed negative symptoms retrieved from psychometric instruments (BNSS) after the intervention | week 0 (t1), week 8 +/- 1 day (t2), week 15 +/- 2 days (t3)
  BNSS: 5 domains for the negative symptoms are recorded, namely "blunted affect", "alogie", "asociality", "anhedonia" and "avolition". The BNSS also distinguishes between the anticipatory and the consumptive aspects of anhedonia, which are distinct advantages over other questionnaires such as PANSS or SANS (Kirkpatrick 2011, Marder & Kirkpatrick 2014). With its 13 items that can be collected within 15 minutes, the BNSS is a short scale that, despite its shortness, has excellent inter-rater and test-retest reliability and good validity. Furthermore, there are only small correlations of the BNSS with masses of positive symptoms, anxiety and depression (Strauss et al., 2012, Kirkpatrick et al., 2011). Like the PSP scale, the BNSS is surveyed during the first, second and third rounds and here too the surveys are conducted by experienced psychologists or psychiatrists.
Changed psychosocial functioning after the intervention (PSP) | week 0 (t1), week 8 +/- 1 day (t2), week 15 +/- 2 days (t3)
  PSP: External rating scale consisting of 4 subscales, which are calculated to a total score ranging from 0 to 100. The 4 scales are "disturbing and aggressive behavior," "self-care," "socially beneficial activities," and "personal and social relationships" (Morosini et al., 2000). The individual items are queried on a 6-point scale, which includes the expressions "absent", "easy", "obvious", "pronounced", "severe" and "extremely serious". Explanations are available for the respective characteristics. Schaub and Juckel (2011) have also created an interview guide for the German version, which should further simplify the assessment. The individual surveys are carried out by experienced psychologists or psychiatrists. The PSP scale was chosen because it is quick and easy to query, has a higher information content than other scales (e.g., SOFAS or GAF), and also has high validity and reliability.

SECONDARY OUTCOMES:
Changed quality of life (Quality of Life Questionnaire in Schizophrenia (S-QoL) | week 0 (t1), week 8 +/- 1 day (t2), week 15 +/- 2 days (t3)
  This is done using the standardized method S-QoL (Auquier et al., 2003). It uses 41 items to record 8 subscales of the quality of life such as well-being, self-esteem, resilience and autonomy. The S-QoL is a self-assessment tool and its application takes 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Brackmann, Dr. phil., Principal Investigator — University Hospital of Psychiatry Zurich, Department of Forensic Psychiatry
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughlings-Jackson, J. (1931). Selected Writings, Taylor J (ed). London, Hodder & Stoughton
- [Background] Frith CD, Done DJ. Towards a neuropsychology of schizophrenia. Br J Psychiatry. 1988 Oct;153:437-43. doi: 10.1192/bjp.153.4.437. PMID 3074851
- [Background] Calvo P, Fortuny JR, Guzman S, Macias C, Bowen J, Garcia ML, Orejas O, Molins F, Tvarijonaviciute A, Ceron JJ, Bulbena A, Fatjo J. Animal Assisted Therapy (AAT) Program As a Useful Adjunct to Conventional Psychosocial Rehabilitation for Patients with Schizophrenia: Results of a Small-scale Randomized Controlled Trial. Front Psychol. 2016 May 6;7:631. doi: 10.3389/fpsyg.2016.00631. eCollection 2016. PMID 27199859
- [Background] Cerino S, Cirulli F, Chiarotti F, Seripa S. Non conventional psychiatric rehabilitation in schizophrenia using therapeutic riding: the FISE multicentre Pindar project. Ann Ist Super Sanita. 2011;47(4):409-14. doi: 10.4415/ANN_11_04_13. PMID 22194076
- [Background] Barak Y, Savorai O, Mavashev S, Beni A. Animal-assisted therapy for elderly schizophrenic patients: a one-year controlled trial. Am J Geriatr Psychiatry. 2001 Fall;9(4):439-42. PMID 11739071
- [Background] Hajak G, Marienhagen J, Langguth B, Werner S, Binder H, Eichhammer P. High-frequency repetitive transcranial magnetic stimulation in schizophrenia: a combined treatment and neuroimaging study. Psychol Med. 2004 Oct;34(7):1157-63. doi: 10.1017/s0033291704002338. PMID 15697042
- [Background] Holi MM, Eronen M, Toivonen K, Toivonen P, Marttunen M, Naukkarinen H. Left prefrontal repetitive transcranial magnetic stimulation in schizophrenia. Schizophr Bull. 2004;30(2):429-34. doi: 10.1093/oxfordjournals.schbul.a007089. PMID 15279057
- [Background] Jormfeldt H, Carlsson IM. Equine-Assisted Therapeutic Interventions Among Individuals Diagnosed With Schizophrenia. A Systematic Review. Issues Ment Health Nurs. 2018 Aug;39(8):647-656. doi: 10.1080/01612840.2018.1440450. Epub 2018 Mar 6. PMID 29509053
- [Background] Klein E, Kreinin I, Chistyakov A, Koren D, Mecz L, Marmur S, Ben-Shachar D, Feinsod M. Therapeutic efficacy of right prefrontal slow repetitive transcranial magnetic stimulation in major depression: a double-blind controlled study. Arch Gen Psychiatry. 1999 Apr;56(4):315-20. doi: 10.1001/archpsyc.56.4.315. PMID 10197825
- [Background] Kirkpatrick B, Strauss GP, Nguyen L, Fischer BA, Daniel DG, Cienfuegos A, Marder SR. The brief negative symptom scale: psychometric properties. Schizophr Bull. 2011 Mar;37(2):300-5. doi: 10.1093/schbul/sbq059. Epub 2010 Jun 17. PMID 20558531
- [Background] Marder SR, Kirkpatrick B. Defining and measuring negative symptoms of schizophrenia in clinical trials. Eur Neuropsychopharmacol. 2014 May;24(5):737-43. doi: 10.1016/j.euroneuro.2013.10.016. Epub 2013 Nov 11. PMID 24275698
- [Background] Maujean, A., Pepping, C. A., & Kendall, E. (2015). A systematic review of randomized controlled trials of animal-assisted therapy on psychosocial outcomes. Anthrozoös, 28(1), 23-36. doi.org/10.2752/089279315X14129350721812
- [Background] Rollnik JD, Huber TJ, Mogk H, Siggelkow S, Kropp S, Dengler R, Emrich HM, Schneider U. High frequency repetitive transcranial magnetic stimulation (rTMS) of the dorsolateral prefrontal cortex in schizophrenic patients. Neuroreport. 2000 Dec 18;11(18):4013-5. doi: 10.1097/00001756-200012180-00022. PMID 11192620
- [Background] Schaub D, Juckel G. [PSP Scale: German version of the Personal and Social Performance Scale: valid instrument for the assessment of psychosocial functioning in the treatment of schizophrenia]. Nervenarzt. 2011 Sep;82(9):1178-84. doi: 10.1007/s00115-010-3204-4. German. PMID 21174069
- [Background] Villalta-Gil, V., Roca, M., Gonzalez, N., Domenec, E., Cuca, Escanilla, A., ... & Schi-Can group. (2009). Dog-assisted therapy in the treatment of chronic schizophrenia inpatients. Anthrozoös, 22(2), 149- 159. doi.org/10.2752/175303709X434176
- [Background] Andreasen NC. The Scale for the Assessment of Negative Symptoms (SANS): conceptual and theoretical foundations. Br J Psychiatry Suppl. 1989 Nov;(7):49-58. No abstract available. PMID 2695141
- [Background] Auquier P, Simeoni MC, Sapin C, Reine G, Aghababian V, Cramer J, Lancon C. Development and validation of a patient-based health-related quality of life questionnaire in schizophrenia: the S-QoL. Schizophr Res. 2003 Sep 1;63(1-2):137-49. doi: 10.1016/s0920-9964(02)00355-9. PMID 12892868
- [Background] Brenner, H. D., Roder, V., Hodel, B., Kienzle, N., Reed, D., & Liberman, R. P. (1994). Integrated psychological therapy for schizophrenic patients (IPT). Hogrefe & Huber Publishers.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Morosini PL, Magliano L, Brambilla L, Ugolini S, Pioli R. Development, reliability and acceptability of a new version of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) to assess routine social functioning. Acta Psychiatr Scand. 2000 Apr;101(4):323-9. PMID 10782554
- [Background] Strauss GP, Keller WR, Buchanan RW, Gold JM, Fischer BA, McMahon RP, Catalano LT, Culbreth AJ, Carpenter WT, Kirkpatrick B. Next-generation negative symptom assessment for clinical trials: validation of the Brief Negative Symptom Scale. Schizophr Res. 2012 Dec;142(1-3):88-92. doi: 10.1016/j.schres.2012.10.012. Epub 2012 Nov 3. PMID 23127378